CLINICAL TRIAL: NCT01985854
Title: Conversion From Total Intravenous Anesthesia Technique to Desflurane Anesthesia for Long Duration Neurosurgery: A Pilot Study for Assessment of Recovery Parameters
Brief Title: Conversion From Total Intravenous Anesthesia Technique to Desflurane Anesthesia for Long Duration Neurosurgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tokyo Women's Medical University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Makoto Ozaki, Professor, Tokyo Women's Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIVA DES conversion
Record Dates: First submitted 2013-10-07; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Patients Undergoing Elective Craniotomy
Keywords: Desflurane; Propofol; Total intravenous anesthesia; Neurosurgery
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Propofol target-controlled infusion will be kept 2-4μg /ml plasma concentration throughout procedure.
  Interventions: Drug: Propofol
- Desflurane (Experimental): After taking off the electrophysiological monitoring from the patients, discontinue propofol and start desflurane from 6% (dialed concentration) at flow rate of 4L/min for 2 minutes in desflurane group. When achieve end tidal concentration of 4-5%, decrease the flow rate to 2L/min.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Propofol
  Other Names: Diprivan
  Arms: Propofol
Drug: Desflurane
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
Since neurological testing during neurosurgery, such as somato-sensory evoked potentials, motor-evoked potentials, auditory evoked potentials and visual evoked potentials are well maintained their wave-form reactivity with total intravenous anaesthesia technique better than inhalational anesthetic techniques, the standard anesthesia method for neurosurgery is usually total intravenous anaesthesia technique. Nonetheless, after finishing recording the evoked potential responses during surgery, facilitation of recovery from general anesthesia is getting important, because the real neurological physical examination is much more sensitive than above electrical evoked potentials to evaluate the results of surgical operation.

We propose to evaluate the recovery parameters after conversion from total intravenous anaesthesia technique to Desflurane anesthesia during long term neurosurgery procedures. The conversion will be initiated upon completion of the neurophysiological electric evoked potentials assessment. Based on the pharmacological properties of desflurane, we hypothesize that recovery after conversion to Desflurane will be faster compared to recovery after total intravenous anaesthesia alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective craniotomy
* American Society of Anesthesiology Physical Status Ⅰ, II and III
* Age: between 20 to 65 years
* Sex: male or female
* Patients who are postmenopausal or surgically sterilized
* Expected Operation time is longer than 4 hours.

Exclusion Criteria:

-

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time from the discontinuation of anesthesia to extubation | Patients will be followed in the operation room, an expected average of 30 minutes.

SECONDARY OUTCOMES:
Time from the discontinuation of anesthesia to eye opening | At the end of surgery, duration time from the discontinuation of anesthesia to the eye opening will be measured, averaged expected time is 30 minutes
Cognitive function | Up to 24 hours
  Cognitive function will be measured by Mini-Mental state examination at baseline (preoperatively) 5 minutes and 24 hours after extubation. Postoperative recovery function will be also measured by Post-operative Quality Recovery Scale (PQRS scale) at 5 minutes and 24 hours after extubation.
Time from the discontinuation of anesthesia to orientation | Up to 24 hours
  Time from the discontinuation of anesthesia to orientation (State name, state the date of birth)

OTHER OUTCOMES:
Length of ICU stay | Patients will be followed for the duration of intensive care unit stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Ozaki, Ph.D, Study Chair — Tokyo Women's Mecical University, Department of Anesthesiology
Locations (1):
- Tokyo Women's Medical University Hospital, Tokyo, Tokyo, Japan